CLINICAL TRIAL: NCT02246790
Title: Surgical Ablation of Long-standing Persistent Atrial Fibrillation During CABG Through Continuous Subcutaneous Monitoring
Brief Title: Surgical Ablation of Long-standing Persistent AF During CABG
Acronym: LABARFA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Alexander Romanov, Meshalkin Research Institute of Pathology of Circulation, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LABARFA
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: ablation, CABG; Long-standing persistent Atrial Fibrillation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biatrial radiofrequency ablation and CABG (Active Comparator): Biatrial radiofrequency ablation during CABG
  Interventions: Procedure: Biatrial radiofrequency ablation and CABG
- Left atrial radiofrequency ablation and CABG (Active Comparator): Left atrial radiofrequency ablation during CABG
  Interventions: Procedure: Left atrial radiofrequency ablation and CABG

INTERVENTIONS:
Procedure: Biatrial radiofrequency ablation and CABG — Coronary artery bypass (CABG) using cardio-pulmonary bypass (CPB) and occlusion. Concomitant biatrial RFA during CPB.
  Arms: Biatrial radiofrequency ablation and CABG
Procedure: Left atrial radiofrequency ablation and CABG — Coronary artery bypass (CABG) using cardio-pulmonary bypass (CPB) and occlusion. Concomitant left atrial RFA during CPB.
  Arms: Left atrial radiofrequency ablation and CABG

SUMMARY:
Purpose. Comparison of outcomes in patients underwent CABG combined with left atrial and biatrial radiofrequency ablation of long-standing persistent atrial fibrillation.

Hypothesis of the study - patients with long-standing persistent atrial fibrillation and coronary artery disease after CABG in combination with biatrial RFA have a better outcomes for the freedom of AF compared with patients undergoing left atrial RFA during CABG.

DETAILED DESCRIPTION:
This is a single blinded prospective randomized study involving 116 patients with long-standing persistent AF and coronary artery disease. 116 patients are required to have a 80% chance of detecting, as significant at the 5% level, an increase in the primary outcome (freedom fro AF) measure by 12% in the biatrial group over left atrial group. Patients are divided into two groups, group I - biatrial + CABG (58 patients), and group II - left atrial + CABG (58 patients). Randomization is conducted by using accidental sampling before operation. The blinding process is applied to a patient, who is informed about received coronary artery bypass grafting, but don't know about kind of surgical ablation. Subcutaneous cardiac monitor is implanted to all patients for cardiac rhythm monitoring.

ELIGIBILITY:
Inclusion criteria:

* American College of Cardiology (ACC)/ American Heart Association (AHA) Indications for CABG
* At least 2 ECG-verified (12-channel ECG, Holter telemetry) long-term persistent AF within last 12 months
* The patient's consent to participate in the study

Exclusion Criteria:

* Intolerance of antiarrhythmic drugs
* Heart valve disease requiring invasive treatment
* Left atria more than 6.5 cm
* Prior cardiac surgery
* Active pacemaker treatment
* Active anti-arrhythmic treatment (AAD) class I and III
* Contraindication to oral anticoagulant/heparin treatment
* Ejection fraction less than 30 % (EF < 30 %) assessed by transthoracic echocardiography

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation | up to 36 months
  Freedom from AF. All cases of AF after surgical intervention.
  Atrial fibrillation is defined as atrial fibrillation paroxysm lasting at least 60 seconds. Patients with AF>0.5% were classified as non-responders.

SECONDARY OUTCOMES:
Cardiovascular events | Within three years after surgery
  All cases of stroke, cardiac infarction, thromboembolism, bleeding and death

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin State Research Institute of Circulation Pathology, Novosibirsk, Russia